CLINICAL TRIAL: NCT05616520
Title: Clinical Efficacy for the Treatment of Complex Femoropopliteal Artery Lesions Using Drug-coated PTA Balloon：a Real-world Registry Study(CARPLAY-DCB Study)
Brief Title: Treatment of Complex Femoropopliteal Artery Lesions Using Drug-coated PTA Balloon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Changhai Hospital (Other); Tianjin Medical University General Hospital (Other); Second Affiliated Hospital of Suzhou University (Other); Fudan University (Other); RenJi Hospital (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital of Zhejiang University (Other); Chengdu University of Traditional Chinese Medicine (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CARPLAY-DCB Study
Record Dates: First submitted 2022-09-01; First posted 2022-11-15 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-06

CONDITIONS: Peripheral Arterial Disease
Keywords: drug-coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: drug-coated balloon — The intervention relates to a drug-coated balloon catheter includes a balloon and cover the drug-coated balloon surface.

SUMMARY:
Although DCBs had been widely applicable after registration, there are still lack of clinical data and evidence in the real world condition of Chinese population. This data collection aims to perform regularly clinical follow up to guide the standardized diagnosis and treatment of patients post-operatively, in order to achieve the maximum clinical benefits of these patients, as well as improve the development of the field of peripheral artery disease treated by drug-coated balloon.

DETAILED DESCRIPTION:
Historically, symptomatic PAD was treated with surgical bypass; however endovascular treatment is now the first line treatment when medical therapy fails. Several endovascular treatment options exist including percutaneous transluminal angioplasty (PTA), stenting with bare metal or drug-eluting stents (DES), cutting balloons, atherectomy, laser debulking. Moreover, drug-coated balloon（DCB）has emerged as a potential treatment option, combining acute restoration of vessel patency by balloon dilatation with long term maintenance of such patency by the anti-proliferative drug delivered by the balloon surface. Results from numerous clinical studies with paclitaxel coated balloons have been reported for the safety and efficacy for peripheral artery diseases.

Besides Medtronic IN.PACT Admiral, other DCBs approved for marketing in Chinese Mainland include Acoart (Acotec, China), Reewarm ® PTX (endovastec, China), Ultrafree (ZYLOX, China). Although DCBs had been widely applicable after registration, there are still lack of clinical data and evidence in the real world condition of Chinese population. Therefore, the data collection can also further expand and understand the experience of using DCB in a real world patient population in China, especially for the surveillance of safety events, in order to ensure the long-term application safety in Chinese population. Moreover, this data collection aims to perform regularly clinical follow up to guide the standardized diagnosis and treatment of patients post-operatively, in order to achieve the maximum clinical benefits of these patients, as well as improve the development of the field of peripheral artery disease treated by drug-coated balloon.

ELIGIBILITY:
Inclusion Criteria:

1. Rutherford grade 2-5.
2. Femoropopliteal artery disease (stenosis > 50%) with at least one of following complex lesion characteristics: - long lesion (>150 mm), CTO(>50 mm),in-stent restenosis(Tosaka Ⅱ、Ⅲ), calcified lesion (PACCS grade 2-4)
3. Patients who understand the purpose of this study, volunteer to participate in the experiment, sign informed consent and are willing to follow up.
4. The guidewire needs to pass through the lesion.
5. Life expectancy> 24 months.
6. Patients who received DCB intervention after thrombus removal through PMT or CDT.
7. Patients who have received DCB intervention for both lower limbs can be enrolled in the group according to the intracavitary treatment time.
8. There is at least one continuous below-the-knee outflow artery or obtained by endovascular reconstruction.
9. For patients combined aortic iliac artery disease, the inflow can be recanalized after endovascular reconstruction without illiac residual stenosis exceeding 50%.

Exclusion Criteria:

1. Patients with stroke, cerebral hemorrhage, gastrointestinal hemorrhage or myocardial infarction within 3 months before enrollment.
2. Patients who are known to be allergic to heparin, aspirin, other antiplatelet drugs, contrast agents, etc.
3. Patients who have participated in clinical trials of drugs or other medical devices that interfere with this clinical trial within the past 3 months.
4. Pregnant and lactating women.
5. Patients who are unable or unwilling to participate in this trial.
6. Patients with Buerger's disease.
7. Patients who have undergone arterial bypass on the treatment side.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with complex femoralpopliteal artery lesions.
Sampling Method: Probability Sample
Enrollment: 838 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from clinically-driven target lesion revascularization(CD-TLR) | 24 months
  Primary patency is defined as freedom from clinically driven TLR and freedom from restenosis as determined by duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) ≤ 2.4

SECONDARY OUTCOMES:
Primary patency | 1 month, 3 months, 6 months, 12 months, 24 months
  Primary patency is defined as freedom from clinically driven TLR and freedom from restenosis as determined by duplex ultrasound (DUS) Peak Systolic Velocity Ratio (PSVR) ≤ 2.4
Freedom from clinically-driven target lesion revascularization(CD-TLR) | 1 month, 3 months, 6 months, 12 months, 24 months
  Clinically-driven target lesion revascularization (CD-TLR) is defined as any re-intervention within the target lesion due to symptoms or drop of ankle brachial index (ABI) of ≥20% or >0.15 when compared to post-procedure baseline.
Major adverse events | 1 month, 3 months, 6 months, 12 months, 24 months
  Operation-related acute thrombosis, arterial embolism, major amputation and all-cause mortality.
Technical success rate | 1 week
  Successfully revascularize the target vessel. The residual stenosis is <30% and there is no acute thrombosis occurred in the target vessel within 1 week post-operation.
Rutherford classification change | 1 month, 3 months, 6 months, 12 months, 24 months
  Rutherford classification change including ulcer healing in patients with Rutherford grade 5
improvement of EQ-5D-5L | 1 month, 3 months, 6 months, 12 months, 24 months
  Improvement in the European Five Dimensional Health Scale (EQ-5D-5L) at 1 month, 3 months, 6 months, 12 months, and 24 months after surgery.
improvement of Vas-QoL | 1 month, 3 months, 6 months, 12 months, 24 months
  Improvement in the quality of life scores (Vas-QoL) at 1 month, 3 months, 6 months, 12 months, 24 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Laird JA, Schneider PA, Jaff MR, Brodmann M, Zeller T, Metzger DC, Krishnan P, Scheinert D, Micari A, Wang H, Masters M, Tepe G. Long-Term Clinical Effectiveness of a Drug-Coated Balloon for the Treatment of Femoropopliteal Lesions. Circ Cardiovasc Interv. 2019 Jun;12(6):e007702. doi: 10.1161/CIRCINTERVENTIONS.118.007702. Epub 2019 Jun 14. PMID 31195825
- [Background] Soga Y, Iida O, Fujihara M, Kawasaki D, Saito S, Urasawa K, Yokoi H, Fernandez EJ, Guo J, Nakamura M; IN.PACT Japan Post-Market Surveillance Study. Real-World Clinical Outcomes of IN.PACT Admiral Drug-Coated Balloon for Femoropopliteal Artery Disease - 12-Month Results From Japan Post-Market Surveillance Study. Circ J. 2021 Nov 25;85(12):2149-2156. doi: 10.1253/circj.CJ-21-0491. Epub 2021 Oct 6. PMID 34615815